CLINICAL TRIAL: NCT06268405
Title: Breast Cancer Combined Visualization And Characterization Tools - Novel Positron Emission Mammography System and Liquid Biopsy
Brief Title: Positron Emission Mammography and Liquid Biopsy in Women With High-risk Breast Screenings
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Radialis Inc. (Industry); The Princess Margaret Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 22-5806
Record Dates: First submitted 2024-02-12; First posted 2024-02-20 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer
Keywords: Positron Emission Mammography (PEM); Liquid Biopsy
MeSH Terms: conditions — Breast Neoplasms | interventions — Liquid Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Liquid Biopsy and Positron Emission Mammography (PEM) (Experimental): To perform the Liquid Biopsy assays, a baseline blood sample will be collected prior to the MRI-guided biopsy, and a follow-up blood and a tissue sample (if available) may be requested post-surgery If malignancy is confirmed by the standard of care histopathology results.
  To perform the Positron Emission Mammography (PEM), participants will be injected with 74 megabecquerel (MBq) of commercially distributed 2-[fluorine-18]-fluoro-2-deoxy-D-glucose (F-18 FDG). Following a delay of one hour for F-18 FDG uptake, the study participants will undergo a bilateral 4-view combination PEM scan.
  Interventions: Genetic: Liquid Biopsy; Device: Positron Emission Mammography (PEM)

INTERVENTIONS:
Genetic: Liquid Biopsy — Detects cell-free DNA (cfDNA) circulating in the blood by whole-genome sequencing (WGS). It also detects cfDNA containing epigenetic marks by cell-free methylated DNA immunoprecipitation and high throughput sequencing assays and may determine the concordance of genomic alterations between tumour tissue (if available) and matched plasma samples by WGS.
Device: Positron Emission Mammography (PEM) — PEM produces high-sensitivity images of breasts with low levels of F-18 FDG.

SUMMARY:
The goal of this research study is to evaluate the performance of two experimental tests, namely Liquid Biopsy and Positron Emission Mammography (PEM) in women at high risk of breast cancer. The plan for this study is to assess whether findings from the combination or each individual test can assist radiologists in visualizing and characterizing beast abnormalities.

Liquid Biopsy is a blood test that can detect early tumours in patients with malignancies, while PEM is an imaging tool equipped with a high-resolution camera that uses a low dose of injected positron emitting isotope to locate breast tumours. Participation in this study entails a blood draw for Liquid Biopsy test and a PEM imaging exam before undergoing a magnetic resonance imaging (MRI) - guided biopsy for a suspicious breast lesion.

If PEM and/or Liquid Biopsy provide accurate information to assist radiologists in visualizing and characterizing breast abnormalities, this method may serve as the first step towards establishing these genomic and new imaging technologies as new diagnostic modalities and ultimately reduce the unnecessary biopsies and anxiety in high-risk populations.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are older than 18 years of age
* Individuals who are planned to undergo an MRI-guided biopsy based on high- risk screening imaging detected lesions
* Individuals with the ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* High-risk Individuals with screening-imaging studies without suspicious lesions detected by the standard of care mammogram and/or MRI
* Individuals who are pregnant or who think they may be pregnant
* Individuals who are breast-feeding
* Individuals with known allergies to F-18 FDG

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-21 (Actual); Primary Completion 2025-09-21 (Estimated); Study Completion 2026-09-21 (Estimated)

PRIMARY OUTCOMES:
Evaluating the performance of PEM and Liquid Biopsy in visualizing and characterizing breast abnormalities | 3 years
  The performance of PEM and/or Liquid Biopsy, including percent sensitivity, specificity, positive and negative predictive values, in visualization and characterization of suspicious breast abnormalities will be evaluated and compared to magnetic resonance imaging (MRI), and digital mammography.

CONTACTS AND LOCATIONS:
Overall Officials: Vivianne Freitas, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada